CLINICAL TRIAL: NCT06346379
Title: The Effect of Baduanjin on Physical Fitness and Bone Density in Maintenance Hemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-K086-01
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-03

CONDITIONS: Rehabilitation; Physical Fitness; Bone Density; Hemodialysis Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin exercise (Experimental): Before starting dialysis, Patients perform Baduanjin exercises. All Baduanjin training is provided by a professional doctor who has received training on BaduanJin and obtained certificate. Each session is approximately 30 minutes in duration, consisting of 5 minutes of warm-up exercises, 20 minutes of Baduanjin practice, and 5 minutes of cool-down exercises.
  Interventions: Behavioral: Baduanjin exercise
- Control group (No Intervention): Patients in this group maintain their conventional therapy and daily life activities, and there is no intervention given.

INTERVENTIONS:
Behavioral: Baduanjin exercise — Baduanjin has 8 movement forms, which are easy to learn without special equipment.These advantages make Baduanjin a suitable exercise for dialysis patients.The movements involved in Baduanjin require the individual to reach beyond the base of support, change the base of support between bilateral and unilateral stance, and perform movements in a sustained squatting posture. These maneuvers challenge balance and require muscle strength to be executed successfully.During the exercise of Baduanjin, the knees are half bent and the body center of gravity is stable between the feet, which can effectively develop the strength and endurance of skeletal muscle groups, improving the physical fitness and Bone mineral density.
  Arms: Baduanjin exercise

SUMMARY:
The aim of this study is to examine the effect of 18-month Baduanjin exercise on physical fitness and bone density in maintenance hemodialysis (MHD) patients. 50 MHD patients aged 18-75 will included in this study and randomly divided into two groups (intervention group and control group). The intervention group will be led by a professional person and underwent Baduanjin exercise three times a week before hemodialysis. The control group maintained routine treatment and daily activities.

DETAILED DESCRIPTION:
The aim of this study is to observe the therapeutic effect of Baduanjin on improving physical fitness and bone density in MHD patients. A total of 50 MHD patients will be included and randomized into an intervention group of 25 cases and a control group of 25 cases. The intervention group undergo a 30 minute Baduanjin exercise under the guidance of a professional doctor before the dialysis day, including a 5-minute warm-up exercise, a 20 minute Baduanjin exercise, and a 5-minute relaxation exercise. The intervention group practice three days a week, while the control group maintain routine treatment and daily activities. Measure the indicators of each group at baseline, months 6, 12,18. The evaluation of physical fitness is based on the scores (which include muscle strength measurement; five-times sit-to-stand test; timed "up and go" test; sitting forward flexion test; standing on one-leg with eyes closed test ). The bone mineral density test is based on the result of the double-energy DXA line. The quality of life score is based on the SF-12 score, and the emotional score is based on the anxiety and depression scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old;
2. Having received MHD treatment in this dialysis center for more than 3 months and maintaining stable condition;
3. Having normal comprehension ability, clear verbal expression, informed consent and willingness to participate in this study.
4. Having free movement ability, and being able to tolerate Baduanjin exercise after cardiopulmonary exercise test;
5. Right-handed, with fistula in the non-dominant hand;

Exclusion Criteria:

1. Patients who usually practice traditional Chinese medicine exercises such as tai chi;
2. Patients who are recently complicated with severe infections, active malignant tumors, severe cardiopulmonary insufficiency, gastrointestinal bleeding, nervous system diseases and cannot tolerate exercise;
3. Patients with various orthopedic, neurological, and other diseases that cause muscle and joint deformities that affect grip strength measurement;
4. Patients with senile dementia, hearing impairment, comprehension abnormalities, mental disorders, unclear verbal expression or unwilling to participate in this study;
5. Patients with hemoglobin <70g/L, carbon dioxide binding capacity <13mmol/L, and blood potassium >6.5mmol/L in laboratory tests and no significant improvement after treatment;
6. Patients who are participating in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle strength measurement | 0 month, 6month, 12month，18month
  Grip strength can reflect the strength of hand muscles. The grip strength of both hands of patients was measured using a domestic gripper.The patient took an upright position and grasped the handle with the maximum force. When the display on the machine stopped changing, the value was recorded. The test was repeated three times, and the maximum value was taken to record the results.
Five-times Sit-to-Stand Test (FTSST) | 0 month, 6month, 12month，18month
  The five-times sit-to-stand test is used to evaluate the functional strength of the lower limbs. MHD patients sat on a 46cm chair without armrests, with their feet on the ground and their backs not resting on the chair. Their hands were crossed on their shoulders. They stood up from the chair as quickly as possible without arm support. They completed five sitting and standing movements, and the completion time was recorded.During the test, the patient kept his hands crossed and his knees completely straightened.Three tests were completed, with a one-minute rest between tests. The average value of the three tests was statistically analyzed.
Timed "up and go" test (TUGT) | 0 month, 6month, 12month，18month
  The timed "up and go" test is often used to evaluate functional mobility such as balance and walking required in daily life.MHD patients were seated in a back chair with armrests (the seat was about 46cm high, and the armrest was about 21cm high). A guide line was placed on the ground 3m away from the chair. After the test began, the patient left the chair, stood firmly and walked forward for 3m as fast as possible, crossed the guide line, turned around, and returned to the chair to sit down. The walking aids were not allowed during the test.The test was conducted 3 times in total, with a 1-minute rest between adjacent tests. The average value of the 3 tests was taken for statistical analysis.
The sitting forward flexion test | 0 month, 6month, 12month，18month
  The sitting forward flexion test is often used to evaluate the flexibility of the lower limbs of patients.The patient straightened the knee joint, sat on the flat ground with both feet flat on the test board, bent forward, straightened both arms forward, and gradually pushed the cursor with both middle fingertips to the farthest possible distance.The measuring device was 0 point along the plane of the foot pedal board, negative inward, positive forward, in centimeters. The knee joint could not be bent during the test, and sudden force could not be applied.The test was conducted 3 times in total, and the best result was taken for statistical analysis.
The Standing on one-leg with eyes closed test (SOLECT) | 0 month, 6month, 12month，18month
  The Standing on one-leg with eyes closed test evaluates the stability of the static posture by quantitative measurement, reflecting the balance ability of patients.The patient spread both hands, closed his eyes, and stood on one leg, with the other leg bent so that the angles between the two legs were 90 degrees. Time was recorded from the time when the foot left the ground, and the shaking stopped when the foot left the ground or stood up. The average of the three times was used for statistical analysis.
Bone mineral density test | 0 month, 6month, 12month，18month
  The signals received by the scanning system after the double-energy DXA line penetrated the body were transmitted to the supporting software to calculate the average bone mineral density content (g/cm2) of the whole body, the left femur Ward triangle area, and the lumbar spine (L2~L4).

SECONDARY OUTCOMES:
Changes in the Short Form-36(SF-36) | 0 month, 6month, 12month，18month
  Changes from the Short Form-36 (SF-36) and European Quality of Life Five Dimension（EQ-5D-5L）scale at 0 months, 6 months, 12 months. The SF-36 score is used to evaluate an individual's health status and quality of life. The SF-36 score expressed as a number between 0 and 100, with higher numbers indicating better health.
Changes in the Hospital Anxiety and Depression Scale （HADS） | 0 month, 6month, 12month，18month
  Changes from HADS Index at at 0 months, 6 months, 12 months. HADS consists of 14 items, of which 7 items assess depression and 7 items assess anxiety. The scores for anxiety and depression range from 0 to 21, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yuan, Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Data can be shared after request

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06346379/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06346379/ICF_001.pdf